CLINICAL TRIAL: NCT03532906
Title: Is it Feasible to Conduct a Randomised Controlled Trial (RCT) of the Transverse Abdominis Plane (TAP) Block Versus Anaesthetic Injections to the Wound Site for Patients Requiring Laparoscopic Cholecystectomy?
Brief Title: Feasibility Study on Pain Control After Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 1901750
Record Dates: First submitted 2018-04-27; First posted 2018-05-22 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-03

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAP block (Active Comparator): Patients receive the injection of local anaesthetic into the right abdominal wall (TAP block) together with the injection of local anaesthetic into the surgical wounds.
  Interventions: Drug: TAP Block
- Control (Other): Patients receive the injection of local anaesthetic into the surgical wounds only.
  Interventions: Drug: Control

INTERVENTIONS:
Drug: TAP Block — Injection of Bupivacaine 0.5% 20 ml into the thickness of the right abdominal wall and of Bupivacaine 0.5% 10 ml into the surgical wounds.
  Other Names: Bupivacaine 0.5%
  Arms: TAP block
Drug: Control — Injection of Bupivacaine 0.5% 10 ml into the surgical wounds
  Other Names: Bupivacaine 0.5%
  Arms: Control

SUMMARY:
The objective of the study is to hopefully understand the most beneficial way to control pain after removing the gallbladder by keyhole surgery (laparoscopic cholecystectomy).

The investigators will investigate two groups of patients undergoing laparoscopic cholecystectomy.

One group will receive the injection of local anaesthetic into the abdominal wall (TAP block) and into the wounds; the second group will have local anaesthetic into the wounds only.

In order to have meaningful results, we anticipate a large number of participants would be required. Therefore we would test first whether it is technically possible to set up the study itself.

The investigators will be looking at parameters (willingness of patients to be recruited, willingness of clinicians to recruit participants, number of eligible patients, follow-up rates, adherence/compliance rates, number of participants needed for an adequate sample size) that will allow to understand if such a larger trial is technically possible to set up.

DETAILED DESCRIPTION:
Pain control after laparoscopic cholecystectomy can be achieved with the injection of local anaesthetic into the abdominal wall (TAP block) or into the surgical wounds. There is no reported literature comparing the two techniques with regard to early discharge rate, consumption of oral painkillers and return to daily activities in the week following surgery. In an era where day case surgery has become reality, there is a pressing need for strategies to optimize patients' pathways. In this context the postoperative pain control is a key point.

To compare the two techniques in a randomized trial, a large number of participants would be needed. Therefore the investigators would conduct a pilot study first, to evaluate if further research in the form of a larger study is likely to demonstrate the benefits of the TAP block during laparoscopic cholecystectomy.

During the developing of the research proposal, advice and comments had been given by the local Research and Development Department and the public.

Recruitment

Clinicians will identify potential participants in the surgical outpatient clinic. All patients who fulfil the entry criteria will be invited to take part in the study.

Participants will be fully informed verbally about the proposed study and will receive a Letter of invitation to participant and a Patient information leaflet to take home. That will give them adequate time to read the documents and make an informed choice.

Sample size

As being a feasibility study it is required to have 30 cases per group in the final dataset, with a total of 60 patients.

Consent

Patients will be informed about the study and receive the information leaflet at the time they are enrolled for an elective laparoscopic cholecystectomy in the surgical outpatient clinic. Only once patients are fully informed will they be asked to make a decision to enter the trial. Participants willing to join the study will have written informed consent, on the day of surgery.

Patients will be informed that they do not have to take part in the study if they choose to not be enrolled. Refusal to enter the trial will not compromise their care. Patients will also be informed that if at any time during the study they wish to withdraw they can do so, without having to give a reason and again this will not compromise their care. General Pratictioners will be informed by letter of their patients' inclusion in the study.

Risks and Benefits

There are no additional risks over and above participants' normal clinical care.

Both anaesthetic techniques are currently in use in the Royal Devon and Exeter National Heath System Foundation Trust. The procedures themselves do have potential risks (side-effects) which would be explained routinely to both trial and non-trial patients ahead of surgery. Taking part in this study will not change these risks in any way.

There are no immediate benefits to the participants from taking part in the trial at present. However, if the results are promising, the investigators will run a larger trial that could potentially lead to a new way of looking after patients having laparoscopic cholecystectomy.

That may therefore lead to a future change in medical care that could help patients who will be having laparoscopic cholecystectomy.

The investigators would be clear that no new technique or medication is being tested. Also there is no financial benefit from the study to both the participants and the research team.

Conflicts of Interest

None.

Confidentiality

All data will be stored anonymously against a participant number. Only the clinical team and research nurse will have access to the single table correlating participant's name number. Anonymity will be preserved throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients able/willing to give informed consent for participation in the study.
* Male or female aged 18-60 years old.

Exclusion Criteria:

* Patients having an open cholecystectomy (performed through the standard "rope" incision).
* Patients intended to have laparoscopic cholecystectomy as an inpatient (staying overnight after surgery).
* Patients initially scheduled to have day case surgery but eventually admitted to hospital due to surgical or anaesthetic concerns or social reasons.
* Patients with contraindications in having injection of the local anaesthetic used in the study (i.e. history of side-effects, allergy).
* Patients who cannot have one or more standard oral painkillers prescribed postoperatively.
* Patients with history of chronic pain who are already on long term painkillers.
* Patients unable/unwilling to give informed consent for participation in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-04-26 (Actual)

PRIMARY OUTCOMES:
Total amount number of patients who give their consent to take part to the study | 24 months
  Overall ability to recruit participants
Total number of questionnaire responses | 24 months
  Ability to follow-up participants
Total number of number of patients adhering to follow-up | 24 months
  Ability to collect adequate data

SECONDARY OUTCOMES:
Standard deviation (SD) of hospital stay between the two study arms | 24 months
  To understand if the intervention significantly impacts the length of hospital stay
Standard deviation (SD) of questionnaire scores between the two study arms | 24 months
  To understand if the intervention significantly impacts the scores on the follow-up questionnaire
Standard deviation (SD) of costs (hospital stay and prescription of painkillers) between the two study arms | 24 months
  To understand if the intervention significantly yields a financial benefit

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Manzelli, MD, PhD, Principal Investigator — Royal Devon and Exeter NHS Foundation Trust
Locations (1):
- Royal Devon and Exeter NHS Foundation Trust, Exeter, United Kingdom

IPD SHARING:
Plan to Share IPD: No
It is a feasibility study therefore sharing of individual participant data is not considered for further studies.

REFERENCES:
- [Result] Rafi AN. Abdominal field block: a new approach via the lumbar triangle. Anaesthesia. 2001 Oct;56(10):1024-6. doi: 10.1046/j.1365-2044.2001.02279-40.x. No abstract available. PMID 11576144
- [Result] Baeriswyl M, Kirkham KR, Kern C, Albrecht E. The Analgesic Efficacy of Ultrasound-Guided Transversus Abdominis Plane Block in Adult Patients: A Meta-Analysis. Anesth Analg. 2015 Dec;121(6):1640-54. doi: 10.1213/ANE.0000000000000967. PMID 26397443
- [Result] Charlton S, Cyna AM, Middleton P, Griffiths JD. Perioperative transversus abdominis plane (TAP) blocks for analgesia after abdominal surgery. Cochrane Database Syst Rev. 2010 Dec 8;(12):CD007705. doi: 10.1002/14651858.CD007705.pub2. PMID 21154380
- [Result] Siddiqui MR, Sajid MS, Uncles DR, Cheek L, Baig MK. A meta-analysis on the clinical effectiveness of transversus abdominis plane block. J Clin Anesth. 2011 Feb;23(1):7-14. doi: 10.1016/j.jclinane.2010.05.008. PMID 21296242
- [Result] De Oliveira GS Jr, Castro-Alves LJ, Nader A, Kendall MC, McCarthy RJ. Transversus abdominis plane block to ameliorate postoperative pain outcomes after laparoscopic surgery: a meta-analysis of randomized controlled trials. Anesth Analg. 2014 Feb;118(2):454-463. doi: 10.1213/ANE.0000000000000066. PMID 24445643
- [Result] Pourseidi B, Khorram-Manesh A. Effect of intercostals neural blockade with Marcaine (bupivacaine) on postoperative pain after laparoscopic cholecystectomy. Surg Endosc. 2007 Sep;21(9):1557-9. doi: 10.1007/s00464-006-9181-9. Epub 2007 Mar 7. PMID 17342558
- [Result] El-Dawlatly AA, Turkistani A, Kettner SC, Machata AM, Delvi MB, Thallaj A, Kapral S, Marhofer P. Ultrasound-guided transversus abdominis plane block: description of a new technique and comparison with conventional systemic analgesia during laparoscopic cholecystectomy. Br J Anaesth. 2009 Jun;102(6):763-7. doi: 10.1093/bja/aep067. Epub 2009 Apr 17. PMID 19376789
- [Result] Chazapis M, Walker EM, Rooms MA, Kamming D, Moonesinghe SR. Measuring quality of recovery-15 after day case surgery. Br J Anaesth. 2016 Feb;116(2):241-8. doi: 10.1093/bja/aev413. PMID 26787793